CLINICAL TRIAL: NCT01101737
Title: Evaluation of a Nurse-led Hypertension Clinic in Two Inner City General Practices: Randomised Controlled Trial
Brief Title: Trial of a Nurse Led Hypertension Clinic in Inner City General Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: St George's, University of London, St George's, University of London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: General Nursing Council 2007
Record Dates: First submitted 2010-04-09; First posted 2010-04-12 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Hypertension
Keywords: Hypertension, clinical trial, nurse-led clinic, primary care
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Patients not invited to the nurse-led clinic will continue with usual GP care
- Nurse-led blood pressure clinic (Experimental): Patients randomly allocated to the intervention will be invited to a specialist nurse-led blood pressure clinic.
  Interventions: Other: Nurse-led blood pressure clinic

INTERVENTIONS:
Other: Nurse-led blood pressure clinic — Blood pressure will be measured according to protocol.For patients with blood pressure above optimal targets, treatment changes will be discussed with the patient, a visiting consultant physician and the patient's GP. If they agree, the GP will intensify anti-hypertensive treatment with monthly follow up by the specialist nurse until BP targets are achieved.
  Arms: Nurse-led blood pressure clinic

SUMMARY:
The investigators will do a trial in two general practices to see if the introduction of a blood pressure clinic staffed by a specialist nurse supported by visiting consultant improves blood pressure control compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with last recorded blood pressure greater or equal to the British Hypertension Society audit standard

Exclusion Criteria:

* Secondary hypertension
* Housebound
* Non-English speaking
* Another major illness likely to dominate pattern of care e.g. advanced cancer, dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure | 6 months
  This will be assessed using two audits of practice records where blood pressure was measured and recorded independently by practice staff

SECONDARY OUTCOMES:
Proportion of patients in each group with final blood pressure below the British Hypertension Society optimal target | 6 months after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Sally Dean, SRN, Principal Investigator — St George's, University of London; Pippa Oakeshott, MD, Study Director — St George's, University of London
Locations (1):
- St George's, University of London, London, United Kingdom

REFERENCES:
- [Derived] Dean SC, Kerry SM, Khong TK, Kerry SR, Oakeshott P. Evaluation of a specialist nurse-led hypertension clinic with consultant backup in two inner city general practices: randomized controlled trial. Fam Pract. 2014 Apr;31(2):172-9. doi: 10.1093/fampra/cmt074. Epub 2013 Dec 19. PMID 24356073